CLINICAL TRIAL: NCT00840567
Title: Acquisition of Skin Biopsies and Blood Samples From Normal Volunteers and Patients With Benign, Inherited Hematologic Diseases for Research Purposes
Brief Title: Skin and Blood Research Samples From Healthy Volunteers and Patients With Hematologic Diseases
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Key samples protocols will be provided by a collaborator and we were not able to produce IPS lines from human fibroblasts.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 08-1409
Record Dates: First submitted 2009-02-09; First posted 2009-02-10 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Anemia, Sickle Cell
Keywords: Stem cells
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Volunteers (Other): To obtain a one time skin sample (4 ml skin punch biopsy) and one time blood sample (1 teaspoon)
  Interventions: Procedure: Skin biopsy; Procedure: Blood draw & sample
- Patients with benign, inherited hematologic disease (Other): To obtain a one time skin sample (4 ml skin punch biopsy) and one time blood sample (1 teaspoon)
  Interventions: Procedure: Skin biopsy; Procedure: Blood draw & sample

INTERVENTIONS:
Procedure: Skin biopsy
Procedure: Blood draw & sample

SUMMARY:
The investigators plan to obtain skin and blood samples from healthy volunteers and patients with a benign, inherited hematologic disease to use for research to use homologous recombination to correct β-globin gene mutations in therapeutically useful cells, like autologous induced pluripotent stem cells from sickle cell anemia patients.

DETAILED DESCRIPTION:
* To obtain skin biopsy samples from normal healthy volunteers and patients with a benign, inherited hematologic disease, such as sickle cell anemia, to create induced pluripotent stem cells. Pluripotency will be confirmed by injecting potential iPS cell lines into immunodeficient mice, assessing the ability of each line to cause cystic teratomas in recipient mice.
* To define the efficiency of homologous recombination in induced pluripotent stem cells derived from skin biopsy samples.
* To define the efficiency of homologous recombination in human embryonic stem cells using NIH-approved cell lines.
* To establish the genetic consequences of the derivation of human induced pluripotent cells in normal controls or patients with benign, inherited, hematologic diseases, by genomic analysis, including whole genome sequencing.
* To establish the genetic consequences of homologous recombination in human induced pluripotent stem cells and embryonic stem cells by genomic analysis, including whole genome sequencing.
* To obtain blood samples to confirm genetic mutations in patients with an inherited hematologic disease (and to confirm no mutations in healthy volunteers).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18.
* No active systemic skin infection at biopsy site.
* No allergy to lidocaine or other local anesthetics

Exclusion Criteria:

ALL PATIENTS

* History of a bleeding disorder, easy bleeding, or bruising.
* Inability or unwillingness to provide informed consent.

SICKLE CELL PATIENTS

* Platelets ≤ 50,000
* INR ≥ 1.5
* Currently bing given intravenous heparin

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Obtain skin biopsy samples from normal healthy volunteers and patients with a benign, inherited hematologic disease to created induced pluripotent stem cells | 1 year
  Only one biopsy but analysis may take one year.

SECONDARY OUTCOMES:
Define the efficiency of homologous recombination in induced pluripotent stem cells derived from skin biopsy samples. | 1 year
  Only one blood draw and biopsy but analysis may take one year.
Define the efficiency of homologous recombination in human embryonic stem cells using NIH-approved cell lines | 1 year
  Only one blood draw and biopsy but analysis may take one year.
Establish the genetic consequences of the derivation of human induced pluripotent cells in normal controls or patients with benign, inherited hematologic diseases, by genomic analysis, including whole genome sequencing | 1 year
  Only one blood draw and biopsy but analysis may take one year.
Obtain blood samples to confirm genetic mutations in patients with an inherited hematologic disease | 1 year
  Only one blood draw but analysis may take one year.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Ley, M.D., Study Chair — Washington Univerisity School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Park IH, Zhao R, West JA, Yabuuchi A, Huo H, Ince TA, Lerou PH, Lensch MW, Daley GQ. Reprogramming of human somatic cells to pluripotency with defined factors. Nature. 2008 Jan 10;451(7175):141-6. doi: 10.1038/nature06534. Epub 2007 Dec 23. PMID 18157115
- [Background] Park IH, Lerou PH, Zhao R, Huo H, Daley GQ. Generation of human-induced pluripotent stem cells. Nat Protoc. 2008;3(7):1180-6. doi: 10.1038/nprot.2008.92. PMID 18600223
- [Background] Maherali N, Ahfeldt T, Rigamonti A, Utikal J, Cowan C, Hochedlinger K. A high-efficiency system for the generation and study of human induced pluripotent stem cells. Cell Stem Cell. 2008 Sep 11;3(3):340-5. doi: 10.1016/j.stem.2008.08.003. PMID 18786420
- [Background] Okita K, Ichisaka T, Yamanaka S. Generation of germline-competent induced pluripotent stem cells. Nature. 2007 Jul 19;448(7151):313-7. doi: 10.1038/nature05934. Epub 2007 Jun 6. PMID 17554338
- [Background] Takahashi K, Tanabe K, Ohnuki M, Narita M, Ichisaka T, Tomoda K, Yamanaka S. Induction of pluripotent stem cells from adult human fibroblasts by defined factors. Cell. 2007 Nov 30;131(5):861-72. doi: 10.1016/j.cell.2007.11.019. PMID 18035408
- [Background] Stadtfeld M, Nagaya M, Utikal J, Weir G, Hochedlinger K. Induced pluripotent stem cells generated without viral integration. Science. 2008 Nov 7;322(5903):945-9. doi: 10.1126/science.1162494. Epub 2008 Sep 25. PMID 18818365
- [Background] Wernig M, Meissner A, Foreman R, Brambrink T, Ku M, Hochedlinger K, Bernstein BE, Jaenisch R. In vitro reprogramming of fibroblasts into a pluripotent ES-cell-like state. Nature. 2007 Jul 19;448(7151):318-24. doi: 10.1038/nature05944. Epub 2007 Jun 6. PMID 17554336
- [Background] Brambrink T, Foreman R, Welstead GG, Lengner CJ, Wernig M, Suh H, Jaenisch R. Sequential expression of pluripotency markers during direct reprogramming of mouse somatic cells. Cell Stem Cell. 2008 Feb 7;2(2):151-9. doi: 10.1016/j.stem.2008.01.004. PMID 18371436
- [Background] Hockemeyer D, Soldner F, Cook EG, Gao Q, Mitalipova M, Jaenisch R. A drug-inducible system for direct reprogramming of human somatic cells to pluripotency. Cell Stem Cell. 2008 Sep 11;3(3):346-353. doi: 10.1016/j.stem.2008.08.014. PMID 18786421
- [Background] Wernig M, Lengner CJ, Hanna J, Lodato MA, Steine E, Foreman R, Staerk J, Markoulaki S, Jaenisch R. A drug-inducible transgenic system for direct reprogramming of multiple somatic cell types. Nat Biotechnol. 2008 Aug;26(8):916-24. doi: 10.1038/nbt1483. Epub 2008 Jul 1. PMID 18594521
- [Background] Wernig M, Meissner A, Cassady JP, Jaenisch R. c-Myc is dispensable for direct reprogramming of mouse fibroblasts. Cell Stem Cell. 2008 Jan 10;2(1):10-2. doi: 10.1016/j.stem.2007.12.001. Epub 2007 Dec 13. No abstract available. PMID 18371415
- [Background] Huangfu D, Osafune K, Maehr R, Guo W, Eijkelenboom A, Chen S, Muhlestein W, Melton DA. Induction of pluripotent stem cells from primary human fibroblasts with only Oct4 and Sox2. Nat Biotechnol. 2008 Nov;26(11):1269-75. doi: 10.1038/nbt.1502. Epub 2008 Oct 12. PMID 18849973
- [Background] Park IH, Arora N, Huo H, Maherali N, Ahfeldt T, Shimamura A, Lensch MW, Cowan C, Hochedlinger K, Daley GQ. Disease-specific induced pluripotent stem cells. Cell. 2008 Sep 5;134(5):877-86. doi: 10.1016/j.cell.2008.07.041. Epub 2008 Aug 7. PMID 18691744
- [Background] Hanna J, Wernig M, Markoulaki S, Sun CW, Meissner A, Cassady JP, Beard C, Brambrink T, Wu LC, Townes TM, Jaenisch R. Treatment of sickle cell anemia mouse model with iPS cells generated from autologous skin. Science. 2007 Dec 21;318(5858):1920-3. doi: 10.1126/science.1152092. Epub 2007 Dec 6. PMID 18063756
- [Background] Kyba M, Perlingeiro RC, Daley GQ. HoxB4 confers definitive lymphoid-myeloid engraftment potential on embryonic stem cell and yolk sac hematopoietic progenitors. Cell. 2002 Apr 5;109(1):29-37. doi: 10.1016/s0092-8674(02)00680-3. PMID 11955444
- [Background] Wang Y, Yates F, Naveiras O, Ernst P, Daley GQ. Embryonic stem cell-derived hematopoietic stem cells. Proc Natl Acad Sci U S A. 2005 Dec 27;102(52):19081-6. doi: 10.1073/pnas.0506127102. Epub 2005 Dec 15. PMID 16357205
- [Background] Okita K, Nakagawa M, Hyenjong H, Ichisaka T, Yamanaka S. Generation of mouse induced pluripotent stem cells without viral vectors. Science. 2008 Nov 7;322(5903):949-53. doi: 10.1126/science.1164270. Epub 2008 Oct 9. PMID 18845712
- [Background] Hotta A, Ellis J. Retroviral vector silencing during iPS cell induction: an epigenetic beacon that signals distinct pluripotent states. J Cell Biochem. 2008 Nov 1;105(4):940-8. doi: 10.1002/jcb.21912. PMID 18773452
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu